CLINICAL TRIAL: NCT01429857
Title: Prognostic Relevance of High-sensitivity Troponin in Patients With Acute Decompensated Heart Failure
Status: Completed | Type: Observational
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Principal Investigator, Christian Ukena, Dr. med. Christian Ukena, University Hospital, Saarland
Other Study IDs: Hom-AHF-Troponin
Record Dates: First submitted 2011-02-01; First posted 2011-09-07 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Heart Failure
Keywords: Troponin concentration in heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the prognostic value of admission high-sensitivity troponin in patients with acute decompensated heart failure.

DETAILED DESCRIPTION:
Patients admitted for acute decompensated heart failure are included in the study. After gaining informed consent, concentrations of high-sensitivity troponin on admission and on discharge are assessed. 6 months after discharged, the incidence of clinical endpoint (mortality of all cause and of cardiovascular cause, hospitalization) is assessed by telephone contact to the patient and/or the physician. The aim of the study is to investigate the prognostic value of high-sensitivity troponin concentration for predicting death and re-hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission for acute cardiac decompensation
* Systolic and / or diastolic heart failure

Exclusion Criteria:

* Myocardial infarction in the last 4 weeks
* Serum creatinine >2.5 mg/dl
* Pulmonary embolism

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Time to cardiovascular death or hospitalization | 6 Months Follow-Up

SECONDARY OUTCOMES:
Time to all cause death or hospitalization | 6 Months Follow-Up

CONTACTS AND LOCATIONS:
Locations (1):
- Innere Medizin III - Kardiologie, Angiologie und Internistische Intensivtherapie, Homburg, Saarland, Germany

REFERENCES:
- [Derived] Poss J, Ukena C, Kindermann I, Ehrlich P, Fuernau G, Ewen S, Mahfoud F, Kriechbaum S, Bohm M, Link A. Angiopoietin-2 and outcome in patients with acute decompensated heart failure. Clin Res Cardiol. 2015 May;104(5):380-7. doi: 10.1007/s00392-014-0787-y. Epub 2014 Nov 19. PMID 25408112